CLINICAL TRIAL: NCT02352246
Title: Effect of High-Intensity Intermittent Exercise on Abdominal Fat Mass in Type 2 Diabetes Postmenopausal Women.
Brief Title: HIIE and Abdominal Fat Mass in DT2 Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratory of metabolic adaptation to exercise under Physiological and Physiopathological conditions (AME2) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0220
Record Dates: First submitted 2015-01-19; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes; Overweight (BMI > 25); Postmenopausal Women
Keywords: intermittent sprinting; abdominal fat mass; type 2 diabetes; postmenopausal women
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight

ARMS (2):
- steady-state exercise (SSE) (Experimental): The aim of our study was to compare the effects of 16-week steady-state exercise (SSE) program with high intensity intermittent exercise (HIIE) program on total abdominal and visceral fat mass in T2D postmenopausal women.
  Interventions: Procedure: Physical activity programs steady-state exercise (SSE) program
- high intensity intermittent exercise (HIIE) (Other): The aim of our study was to compare the effects of 16-week steady-state exercise (SSE) program with high intensity intermittent exercise (HIIE) program on total abdominal and visceral fat mass in T2D postmenopausal women.
  Interventions: Procedure: Physical activity programs high intensity intermittent exercise (HIIE)

INTERVENTIONS:
Procedure: Physical activity programs steady-state exercise (SSE) program — The aim of our study was to compare the effects of 16-week steady-state exercise (SSE) program with high intensity intermittent exercise (HIIE) program on total abdominal and visceral fat mass in T2D postmenopausal women.
  Arms: steady-state exercise (SSE)
Procedure: Physical activity programs high intensity intermittent exercise (HIIE)
  Arms: high intensity intermittent exercise (HIIE)

SUMMARY:
Postmenopausal women, as men, are more prone to central or android obesity. Abdominal fat mass is associated with an increase of cardiovascular diseases (CVD). In type 2 diabetic (T2D) patients, the risk of CVD mortality is more than double compared with that in age-matched subjects.

Most exercise programs designed for weight loss have focused on steady-state exercise (SEE) of around 30 min at a moderate intensity several times a week. Disappointingly, these kinds of exercise programs have led to little or no fat loss (Shaw et al. 2006). Accumulating evidence suggests that high intensity intermittent exercise (HIIE) has the potential to be an effective exercise protocol for reducing fat of overweight individuals, especially at the abdominal level (Boutcher 2011, Kessler 2012). Despite these results, HIIE program has never been used in TD2 postmenopausal women to favor a specific decrease of abdominal fat mass.

The aim of our study was to compare the effects of 16-week steady-state exercise (SSE) program with high intensity intermittent exercise (HIIE) program on total abdominal and visceral fat mass in T2D postmenopausal women.

It is hypothesized that HIIE compared to SSE program would result in significantly greater reductions in total abdominal and visceral fat mass.

DETAILED DESCRIPTION:
Overweight and obesity levels have escalated worldwide, and these trends are occurring in both developed and developing countries. Fat mass and more precisely abdominal fat mass is linked to the development of cardio-vascular diseases (CVD). Postmenopausal women, as men, are more prone to central or android obesity. In type 2 diabetic (T2D) patients, the risk of CVD mortality is more than double compared with that in age-matched subjects.

Most exercise programs designed for weight loss have focused on steady-state exercise (SEE) during at least 30 min, 2 or 3 times a week. Disappointingly, these kinds of exercise programs have led to little or no fat loss (Shaw et al. 2006). Accumulating evidence suggests that high intensity intermittent exercise (HIIE) has the potential to be an effective exercise protocol for reducing fat of overweight individuals, especially at the abdominal level (Boutcher 2011, Kessler 2012). HIIE involves brief high-intensity, anaerobic exercise followed by brief but slightly longer bouts of very low-intensity exercise.

The aim of our study was to compare the effects of 16-week steady-state exercise (SSE) program with high intensity intermittent exercise (HIIE) program on total abdominal and visceral fat mass in T2D postmenopausal women.

30 T2D postmenopausal women will be randomly assigned to SSE (n= 15) or HIIE (n= 15) group. Subjects performed two sessions by week, on bicycle, during 16 weeks.

SSE: For the SSE protocol, each subject performed 40 min at 50% MAP (maximal aerobic power) HIIE: For the HIIE protocol, each subject performed 8 s of sprinting and 12 s of turning the pedals over slowly (between 20 and 30 r.p.m.) for a maximum of 60 repeats a session.

Total body and regional fat content will be measured using dual-energy x-ray absorptiometry (DXA) before and after the intervention (4 months). The contribution of visceral fat to total abdominal fat will be determined from computed tomography (CT).

The effects of HIIE and SSE program on:

* Total fat mass (and appendicular fat mass) (DXA)
* Total fat free mass (and appendicular fat free mass) (DXA)
* Glycemic profile (plasma HbA1c, plasma glucose)
* Lipid profile (TG, HDL, LDL, total cholesterol)
* Food behavior after training (questionnaires)

will also be compared.

Gaussian distribution of the data will be tested by the Kolmogorov-Smirnov test. Data will be presented as mean ± standard deviation (SD). Comparisons between groups will be made with Mann & Whitney U test or ANOVA when appropriate. Relationships between data will be assessed by Pearson correlation. Significance will be accepted at the p<0.05 level. Statistical procedures will be performed using Statistica.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women (55- 82 years)
* T2D
* BMI ≥ 25 and < 40
* able to follow an exercise protocol
* eating behavior and physical activity stable since at least 3 month

Exclusion Criteria:

* - subject not able to perform exercise after medical examination
* subject not able to perform bicycle exercise (pains)
* chronic infection
* use of β-blocker
* medical treatment that could interfere with the different outcome measures
* Hormonal Replacement Therapy (HRT)
* regular consumption of alcohol
* refusal to sign the consent form

Ages: 55 Years to 82 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
loss of abdominal fat mass (g) | at baseline (T0) and after 4 months of training (T4)
  Total abdominal fat mass will be measured in all patients from DXA using the methodology of Martin et Jensen (1991; L1-L2 to pubic rami) before (baseline, T0) and after 4 months of training (T4).

SECONDARY OUTCOMES:
Change from baseline in visceral fat mass (g) | at baseline (T0) and after 4 months of training (T4)
  calculated from computer tomography, Sottier et al. 2013
Change from baseline in total fat mass (g) determined from DXA | at baseline (T0) and after 4 months of training (T4)
  determined from DXA
Change from baseline in total fat free mass (g) determined from DXA | at baseline (T0) and after 4 months of training (T4)
  determined from DXA
Change from baseline in glycemic profile (plasma HbA1c and plasma glucose measurements) | at T0 and after 4 months of training (T4)
  plasma HbA1c and plasma glucose measurements
Change from baseline in lipid profile (plasma TG, HDL, LDL and total cholesterol measurements) | at baseline (T0) and after 4 months of training (T4)
  plasma TG, HDL, LDL and total cholesterol measurements
Change from baseline in food behavior after training (visual analog scale from Flint et al. 2000) | at baseline (T0) and after 4 months of training (T4)
  visual analog scale from Flint et al. 2000

CONTACTS AND LOCATIONS:
Overall Officials: Martine DUCLOS, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France